CLINICAL TRIAL: NCT05887739
Title: Harmonic Ratio in Patients With GLUT1 Deficiency Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Other Study IDs: Gait analysis in GLUT1DS
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: GLUT1DS1; Dystonia; Gait Disorders, Neurologic; Gait Ataxia
MeSH Terms: conditions — Dystonia; Gait Disorders, Neurologic; Gait Ataxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GLUT1DS: Patients affected by GLUT1 deficiency syndrome
  Interventions: Diagnostic Test: Inertial gait analysis
- Healthy controls: Age and sex matched healthy controls
  Interventions: Diagnostic Test: Inertial gait analysis

INTERVENTIONS:
Diagnostic Test: Inertial gait analysis — All groups will be evaluated with inertial gait analysis

SUMMARY:
Glucose transporter deficiency syndrome type 1 (GLUT1DS) is a rare, genetically determined, neurometabolic disorder .

It is estimated that about 90% of affected patients present various pathological gait patterns. Ataxic, spastic, ataxo-spastic, or dystonic walking are the main manifestations described to date.

The kinematic gait analysis with inertial sensors represents a method that is easily applicable in clinical practice, with possible application in numerous neurological syndromes of the pediatric and adult age.

Through the kinematic gait analysis, it will be possible to obtain an accurate characterization of the gait of patients with GLUT1DS. This will allow, in the first place, a better knowledge of locomotor parameters in this rare cohort of patients. Given that kinematic analysis through a wearable sensor is a method that can be easily integrated into daily clinical practice, the data obtained could become prognostic biomarkers and significant outcome measures of the disease (also in relation to possible improvements deriving from treatment with a ketogenic diet or in the context of future pharmacological trials).

DETAILED DESCRIPTION:
Glucose transporter deficiency syndrome type 1 (GLUT1DS) is a rare, genetically determined, neurometabolic disorder. The recently estimated incidence is around 1.65-2.22/100,000. GLUT1 deficiency syndrome is caused by the presence of pathogenic mutations in the SLC2A1 gene, whose haploinsufficiency leads to a reduced availability of glucose in the brain with repercussions on brain function. Ketogenic dietary therapies (KDT) - diets with a high fat content, reduced carbohydrate content and adequate protein content - represent the current standard of treatment for the syndrome: ketone bodies cross the blood-brain barrier and are an alternative energy source for brain metabolism.

It is estimated that about 90% of affected patients present various pathological gait patterns. Ataxic, spastic, ataxo-spastic, or dystonic walking are the main manifestations described to date.

The kinematic gait analysis with inertial sensors represents a method that is easily applicable in clinical practice, with possible application in numerous neurological syndromes of the pediatric and adult age. A single device worn at the lumbar level can accurately measure spatio-temporal parameters of gait. Moreover, with this tool it is possible to assess several Trunk Inertial Indexes. In particular, the Harmonic Ratio (HR), is a representative index of the fluidity and rhythmicity of gait cycle. Along with the largest Lyapunov exponent (LLE), which is a validated method to quantify gait stability in young and old adults, these are reliable parameter to evaluate any gait alterations in the neurological patient.

Through the kinematic gait analysis, it will be possible to obtain an accurate characterization of the gait of patients with GLUT1DS. This will allow, in the first place, a better knowledge of locomotor parameters in this rare cohort of patients. Given that kinematic analysis through a wearable sensor is a method that can be easily integrated into daily clinical practice, the data obtained could become prognostic biomarkers and significant outcome measures of the disease (also in relation to possible improvements deriving from treatment with a ketogenic diet or in the context of future pharmacological trials).

Finally, the identification of a characteristic gait pattern could facilitate the setting up of ad hoc neuromotor rehabilitation activities that are as personalized as possible.

The study therefore has the innovative objective of providing an accurate analysis of the spatio-temporal and kinematic parameters of gait in patients with GLUT1DS, also providing Trunk Inertial Indexes, and to correlate these characteristics with other clinical manifestations of the syndrome, its natural progression, and response to treatment.

- The study is divided into 2 work-packages (WP):

WP1, which represents the core of the present project, is an observational case-control study.

WP2, which represents a pilot sub-study, is a prospective cohort study.

Within WP1, subjects will participate in a single session (V1).

Within WP2, subjects will be followed up with 4 further visits (V2, V3, V4 and V5, respectively), spaced 6 months apart.

Subjects who meet the inclusion criteria will be enrolled and will participate in the study sessions.

Evaluation scheme foreseen:

Patients will undergo four different visits, at four different times:

* First visit (V1): signing of informed consent, collection of clinical-demographic data, anthropometric measurements, compilation of ABC-Movement 2, instrumental gait analysis.
* Second visit (V2): six months after the previous one, clinical re-evaluation, collection of anthropometric measurements, compilation of ABC-Movement 2, instrumental gait analysis.
* Third visit (V3): six months after the previous one, clinical re-evaluation, collection of anthropometric measurements, compilation of ABC-Movement 2, instrumental gait analysis.
* Fourth visit (V4): six months after the previous one, clinical re-evaluation, collection of anthropometric measurements, compilation of ABC-Movement 2, instrumental gait analysis.
* Fifth visit (V5): six months after the previous one, clinical re-evaluation, collection of anthropometric measurements, compilation of ABC-Movement 2, instrumental gait analysis.

Gait analysis procedure:

To acquire walking data, an inertial sensor (BTS G-Walk, BTS, Milan, Italy) will be placed at the level of the fifth lumbar vertebra (L5) using an ergonomic belt. The inertial sensor communicates with a laptop via Bluetooth connection for data logging and offline analysis. The sensor incorporates a triaxial accelerometer (16 bits/axis), triaxial magnetometer (13 bits), and triaxial gyroscope (16 bits/axis). The sampling frequency is 100 Hz, linear and angular trunk accelerations in the anteroposterior (AP), mediolateral (ML) and vertical (V) directions will be recorded.

The "Walk+" protocol of the G-STUDIO software (G-STUDIO, BTS, Milan, Italy) will be used to detect trunk acceleration, left and right gait cycle phases, and spatiotemporal parameters of pelvic kinematics.

The harmonic ratio will be calculated as trunk acceleration data along three directions (vertical, medio-lateral and anteroposterior), decomposing the components of the signal into its harmonics, as the ratio between the sum of the first 10 even and the first 10 odd harmonic multiples of the fundamental frequencies.

The other Trunk Inertial Indexes calculated will be the largest Lyapunov exponent (LLE), coefficient of variation (CV), log dimensionless jerk score (LDLJ), the recurrence quantification analysis (RQA), as described in a previous work by Castiglia et al. We will also assess the Multiscale entropy (MSE), as described by Bisi et al.

Before the experimental session, participants will receive a thorough explanation of study procedures. Instructions will be given to walk at a speed consistent with the usual walk, along a corridor approximately 3 m wide and 30 m long, in the absence of external factors that may interfere with the cadence and rhythm of the gait cycle. Five consecutive tests will be carried out. The trials will be interrupted if the patient should report intolerance to the procedure, asthenia or pain.

- Statistical Plan:

Referring to the work Castiglia et al 2021, which carries out a kinematic analysis on a cohort of patients with Parkinson's disease vs controls, the investigators hypothesize to obtain a similar effect size of 0.74.

Considering a one-tailed t test for the comparison between the two groups (patients and controls), with alpha significance 0.05 power 0.8 and effect size 0.74, the investigators obtain a minimum number of 24 subjects per group.

A preliminary normality analysis will be performed to decide whether to use parametric or non-parametric methods, through graphical representation and Shapiro Wilk test. Numerical variables will be described as mean and standard deviation (or median and quartiles if appropriate), categorical variables as raw number and percentage.

The two groups will be compared by t test or Mann Whitney for independent samples.

Correlation with age will be verified by Pearson (or Spearman if appropriate) correlation coefficient, both intra-group and globally.

The correlation with the quantitative parameters will be verified by Pearson's (or Spearman's if appropriate) correlation coefficient, both intra-group and globally.

Correlations with qualitative parameters will be evaluated by t test or ANOVA (Mann Whitney or Kruskal Wallis if not normal).

The comparison of HR between V1, V2, V3, V4 and V5 will be performed by repeated measures ANOVA (between group factor, whithin factor at time point).

ELIGIBILITY:
Patients eligibility criteria

Inclusion Criteria:

* Pediatric and adult patients (range 3-60 years) diagnosed with GLUT1 deficiency syndrome according to the recommendations of the International Study Group (Klepper et al., 2020)
* Ability to walk independently the necessary route
* Compliance with study procedures

Exclusion Criteria:

* Presence of other neurological or orthopedic comorbidities that may influence gait assessment
* Poor compliance with study procedures

Healthy controls eligibility criteria:

Inclusion Criteria:

* Typically developing healthy volunteers
* Age range 3-60 years

Exclusion criteria:

* Presence of neurological or orthopedic comorbidities that may influence gait assessment

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients affected by GLUT1 deficiency syndromes will be enrolled by attending our clinic at the IRCCS Mondino Foundation.
  Healthy controls will be age and sex matched people among relatives and caregivers of the patients attending our clinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Harmonic Ratio between patients and healthy controls at baseline | Single evaluation at baseline (V1)
  The primary outcome will be the difference in Harmonic Ratio (HR - continuous variable, without unit of measurement) between patients and healthy controls at baseline
Comparison of largest Lyapunov exponent between patients and healthy controls at baseline | Single evaluation at baseline (V1)
  A co-primary outcome will be the difference in largest Lyapunov exponent (LLE - continuous variable, without unit of measurement) between patients and healthy controls at baseline

SECONDARY OUTCOMES:
Comparison of coefficient of variation between patients and healthy controls at baseline | Single evaluation at baseline (V1)
  A secondary outcome will be the difference in coefficient of variation (CV - continuous variable, without unit of measurement) between patients and healthy controls at baseline
Comparison of normalized jerk score between patients and healthy controls at baseline | Single evaluation at baseline (V1)
  A secondary outcome will be the difference in log dimensionless jerk score (LDLJ - continuous variable, without unit of measurement) between patients and healthy controls at baseline
Comparison of recurrence quantification analysis between patients and healthy controls at baseline | Single evaluation at baseline (V1)
  A secondary outcome will be the difference in recurrence quantification analysis (RQA - continuous variable, without unit of measurement) between patients and healthy controls at baseline
Comparison of Multiscale entropy between patients and healthy controls at baseline | Single evaluation at baseline (V1)
  A secondary outcome will be the difference in Multiscale entropy (MSE - continuous variable, without unit of measurement) between patients and healthy controls at baseline
Comparison of Harmonic Ratio in patients between subsequent visits | Change from baseline (V1) to 6 months after (V2) to 12 months after (V3) to 18 months after (V4) to 24 months after (V5)
  A secondary outcome will be the difference in Harmonic Ratio in patients between the baseline and subsequent visits
Comparison of coefficient of variation in patients between subsequent visits | Change from baseline (V1) to 6 months after (V2) to 12 months after (V3) to 18 months after (V4) to 24 months after (V5)
  A secondary outcome will be the difference in coefficient of variation in patients between the baseline and subsequent visits
Comparison of normalized jerk score in patients between subsequent visits | Change from baseline (V1) to 6 months after (V2) to 12 months after (V3) to 18 months after (V4) to 24 months after (V5)
  A secondary outcome will be the difference in log dimensionless jerk score in patients between the baseline and subsequent visits
Comparison of largest Lyapunov exponent in patients between subsequent visits | Change from baseline (V1) to 6 months after (V2) to 12 months after (V3) to 18 months after (V4) to 24 months after (V5)
  A secondary outcome will be the difference in largest Lyapunov exponent in patients between the baseline and subsequent visits
Comparison of recurrence quantification analysis in patients between subsequent visits | Change from baseline (V1) to 6 months after (V2) to 12 months after (V3) to 18 months after (V4) to 24 months after (V5)
  A secondary outcome will be the difference in recurrence quantification analysis in patients between the baseline and subsequent visits
Comparison of Multiscale entropy in patients between subsequent visits | Change from baseline (V1) to 6 months after (V2) to 12 months after (V3) to 18 months after (V4) to 24 months after (V5)
  A secondary outcome will be the difference in Multiscale entropy in patients between the baseline and subsequent visits

CONTACTS AND LOCATIONS:
Overall Officials: Roberto De Icco, Principal Investigator — IRCCS, Mondino Foundation; Valentina De Giorgis, Principal Investigator — IRCCS, Mondino Foundation
Locations (2):
- Italy (2):
  - Child and Adolescent Epileptology Center, Pavia
  - Headache Science & Neurorehabilitation Center, Pavia

REFERENCES:
- [Background] Alter AS, Engelstad K, Hinton VJ, Montes J, Pearson TS, Akman CI, De Vivo DC. Long-term clinical course of Glut1 deficiency syndrome. J Child Neurol. 2015 Feb;30(2):160-9. doi: 10.1177/0883073814531822. Epub 2014 Apr 30. PMID 24789115
- [Background] Bisi MC, Di Marco R, Ragona F, Darra F, Vecchi M, Masiero S, Del Felice A, Stagni R. Quantitative Characterization of Motor Control during Gait in Dravet Syndrome Using Wearable Sensors: A Preliminary Study. Sensors (Basel). 2022 Mar 10;22(6):2140. doi: 10.3390/s22062140. PMID 35336311
- [Background] Blumenschine M, Montes J, Rao AK, Engelstad K, De Vivo DC. Analysis of Gait Disturbance in Glut 1 Deficiency Syndrome. J Child Neurol. 2016 Nov;31(13):1483-1488. doi: 10.1177/0883073816661662. Epub 2016 Aug 10. PMID 27511993
- [Background] Castiglia SF, Tatarelli A, Trabassi D, De Icco R, Grillo V, Ranavolo A, Varrecchia T, Magnifica F, Di Lenola D, Coppola G, Ferrari D, Denaro A, Tassorelli C, Serrao M. Ability of a Set of Trunk Inertial Indexes of Gait to Identify Gait Instability and Recurrent Fallers in Parkinson's Disease. Sensors (Basel). 2021 May 15;21(10):3449. doi: 10.3390/s21103449. PMID 34063468
- [Background] Castiglia SF, Trabassi D, Tatarelli A, Ranavolo A, Varrecchia T, Fiori L, Di Lenola D, Cioffi E, Raju M, Coppola G, Caliandro P, Casali C, Serrao M. Identification of Gait Unbalance and Fallers Among Subjects with Cerebellar Ataxia by a Set of Trunk Acceleration-Derived Indices of Gait. Cerebellum. 2023 Feb;22(1):46-58. doi: 10.1007/s12311-021-01361-5. Epub 2022 Jan 26. PMID 35079958
- [Background] Castiglia SF, Trabassi D, De Icco R, Tatarelli A, Avenali M, Corrado M, Grillo V, Coppola G, Denaro A, Tassorelli C, Serrao M. Harmonic ratio is the most responsive trunk-acceleration derived gait index to rehabilitation in people with Parkinson's disease at moderate disease stages. Gait Posture. 2022 Sep;97:152-158. doi: 10.1016/j.gaitpost.2022.07.235. Epub 2022 Jul 21. PMID 35961132
- [Background] De Giorgis V, Varesio C, Baldassari C, Piazza E, Olivotto S, Macasaet J, Balottin U, Veggiotti P. Atypical Manifestations in Glut1 Deficiency Syndrome. J Child Neurol. 2016 Aug;31(9):1174-80. doi: 10.1177/0883073816650033. Epub 2016 Jun 1. PMID 27250207
- [Background] Klepper J, Leiendecker B. GLUT1 deficiency syndrome--2007 update. Dev Med Child Neurol. 2007 Sep;49(9):707-16. doi: 10.1111/j.1469-8749.2007.00707.x. PMID 17718830
- [Background] Klepper J, Akman C, Armeno M, Auvin S, Cervenka M, Cross HJ, De Giorgis V, Della Marina A, Engelstad K, Heussinger N, Kossoff EH, Leen WG, Leiendecker B, Monani UR, Oguni H, Neal E, Pascual JM, Pearson TS, Pons R, Scheffer IE, Veggiotti P, Willemsen M, Zuberi SM, De Vivo DC. Glut1 Deficiency Syndrome (Glut1DS): State of the art in 2020 and recommendations of the international Glut1DS study group. Epilepsia Open. 2020 Aug 13;5(3):354-365. doi: 10.1002/epi4.12414. eCollection 2020 Sep. PMID 32913944
- [Background] Pearson TS, Akman C, Hinton VJ, Engelstad K, De Vivo DC. Phenotypic spectrum of glucose transporter type 1 deficiency syndrome (Glut1 DS). Curr Neurol Neurosci Rep. 2013 Apr;13(4):342. doi: 10.1007/s11910-013-0342-7. PMID 23443458
- [Background] Suzuki T, Ito Y, Ito T, Kidokoro H, Noritake K, Hattori A, Nabatame S, Natsume J. Quantitative Three-Dimensional Gait Evaluation in Patients With Glucose Transporter 1 Deficiency Syndrome. Pediatr Neurol. 2022 Jul;132:23-26. doi: 10.1016/j.pediatrneurol.2022.04.012. Epub 2022 Apr 29. PMID 35605310
- [Background] Mehdizadeh S. The largest Lyapunov exponent of gait in young and elderly individuals: A systematic review. Gait Posture. 2018 Feb;60:241-250. doi: 10.1016/j.gaitpost.2017.12.016. Epub 2017 Dec 16. PMID 29304432